CLINICAL TRIAL: NCT06501846
Title: Pipelle® Under Ultrasound Guidance (PUG) to Investigate Post-menopausal Bleeding: Randomised Controlled Trial.
Brief Title: Pipelle® Under Ultrasound Guidance (PUG) to Investigate Post-menopausal Bleeding.
Acronym: PUG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24QC8699
Record Dates: First submitted 2024-06-28; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Cancer; Post-Menopausal Bleeding; Endometrial Hyperplasia
Keywords: Pipelle Endometrial Biopsy; Ultrasound Guidance
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blind Endometrial Biopsy (Placebo Comparator): A Pipelle® endometrial biopsy performed in the routine manner without ultrasound guidance.
  Interventions: Procedure: Pipelle® endometrial biopsy performed without ultrasound guidance
- Ultrasound Guided Endometrial Biopsy (Experimental): A Pipelle® endometrial biopsy performed with transabdominal ultrasound guidance.
  Interventions: Procedure: Pipelle® endometrial biopsy performed under transabdominal ultrasound guidance

INTERVENTIONS:
Procedure: Pipelle® endometrial biopsy performed under transabdominal ultrasound guidance — The placement of an ultrasound probe on the lower abdomen while a Pipelle® endometrial biopsy is obtained.
  Arms: Ultrasound Guided Endometrial Biopsy
Procedure: Pipelle® endometrial biopsy performed without ultrasound guidance — A Pipelle® endometrial biopsy is performed by using touch alone.
  Arms: Blind Endometrial Biopsy

SUMMARY:
TITLE Pipelle® under Ultrasound Guidance (PUG) to investigate post-menopausal bleeding: Randomised Controlled Trial

BACKGROUND Women who are suspected of having endometrial cancer (cancer of the inner lining of the womb) due to vaginal bleeding after the menopause must have a tissue sample taken from this area to determine whether there is an abnormality.

One method of doing this is by using a small biopsy device (such as a Pipelle®) in the outpatient setting. This is referred to as an outpatient endometrial biopsy. However, a significant number of attempted endometrial biopsies are unsuccessful in obtaining a sample that is adequate for laboratory (histopathological) assessment. When an adequate sample is not obtained patients must then undergo more invasive testing.

AIM This trial will use an ultrasound probe placed on the lower stomach (transabdominal ultrasound) to try and guide the doctor performing the endometrial biopsy with the aim of increasing the number of adequate samples that are obtained.

The trial will also investigate if this technique is less painful and more acceptable to patients, and if the time taken for patients to receive definitive treatment after their biopsy is reduced.

ELIGIBILITY All patients presenting with post-menopausal bleeding who have an endometrial thickness of 5mm or above without a contraindication to an outpatient endometrial biopsy.

DESIGN Prospective randomised controlled trial enrolling 92 patients. When patients are entered into the study they will randomly assigned to one of two groups. One group will have their biopsy performed under transabdominal ultrasound guidance and the other will have the biopsy performed using the traditional 'blind' approach without ultrasound guidance. There will be 46 patients in each group.

DURATION The trial will run for three years. The trial will be performed in the outpatient gynaecological oncology department at Queen Charlotte's and Chelsea Hospital, part of Imperial College Healthcare NHS Trust.

DETAILED DESCRIPTION:
BACKGROUND Uterine cancer is the most common gynaecological cancer in the United Kingdom with approximately 9,400 new cases diagnosed each year, over 95% arising from the endometrium. Almost all endometrial cancers are diagnosed after the menopause, with most being detected after a woman presents with bleeding. Any woman presenting to her general practitioner or accident and emergency department with post-menopausal bleeding in the United Kingdom should receive an urgent two week wait referral to rapid access gynaecology services. At this appointment women will typically undergo a transvaginal ultrasound scan to assess the gynaecological anatomy, in particular the endometrium. If the endometrium is deemed to be thickened, at more than 4 or 5mm depending on local guidance, sampling is required to rule out endometrial cancer or its precursor, endometrial hyperplasia.

There are two well established routes for obtaining an endometrial biopsy. These are 'blind' office endometrial sampling and hysteroscopy. If ultrasound has shown any focal pathology such as an endometrial polyp or a submucosal fibroid, then the patient must undergo hysteroscopy so this can be directly visualised and confidently removed. Whilst a highly effective procedure, its primary drawbacks are higher costs, a larger side-effect profile and potentially greater pain than the alternative, blind office endometrial sampling.

If a patient has a uniformly thickened endometrium without any suspicion of focal endometrial pathology they can undergo blind office sampling of the endometrium. This is performed with a variety of thin, specially designed plastic biopsy devices that obtain the sample via localised trauma and vacuum suction. This procedure is less invasive, quicker and simpler to perform than a hysteroscopy, however it has a higher failure rate with roughly 4 in 10 patient not having an adequate sample obtained. This is due to either the endometrial sampler not being successfully introduced into the endometrial cavity, or when successfully introduced, the sample obtained being inadequate for histopathological assessment. These patients are then committed to a hysteroscopy so their endometrium can be safely assessed.

PROPOSED STUDY It is theorised that by using ultrasound guidance, the failure rate of office endometrial biopsies could be reduced. We propose to test in an adequately sized randomised controlled trial, the hypothesis that Pipelle® (Pipelle de Cornier) endometrial biopsies, performed under transabdominal ultrasound guidance, will have a higher success rate than blind biopsies. Potential benefits to patients of positive findings in this study include a reduced number of investigations, reductions in pain and increases in patient satisfaction, and a reduction in time from presentation to definitive treatment.

STUDY DESIGN This will be a single centre, prospective, non-blinded randomised controlled trial carried out in the outpatient gynaecological oncology department at Queen Charlotte's and Chelsea Hospital, part of Imperial College Healthcare NHS Trust. The trial will be carried out by gynaecology doctors of registrar and consultant grade who are deemed competent in gynaecological ultrasound and endometrial sampling. Both the doctor and patient will be aware of the study arm allocated. The trial will aim to have the same number of participants in each arm. The study arms are: (i) Blind Endometrial Biopsy and (ii) Ultrasound Guided Endometrial Biopsy. 92 patients will be enrolled, with 46 in each arm.

Once randomised and ready for an endometrial biopsy to be performed, those allocated to the intervention arm will have a transabdominal ultrasound performed by another gynaecologist in the research team while the Pipelle® biopsy is performed. During the procedure, the research doctor will, to the best of their ability, ensure the Pipelle® is introduced to the level of the fundus and that a sample representative of the endometrium is obtained.

As the patient leaves the clinic room, they will be asked to completed a printed Visual Analogue Scale questionnaire to assess anxiety, pain during and after the procedure, and overall patient satisfaction.

The study endpoint will be whichever is the later of: (i) the histopathology for the final participant being reported with an appropriate management plan made, or (ii) when the final patient has an attempted Pipelle® endometrial biopsy if this was a failed attempt.

DATA COLLECTION Demographic patient data collected will include age, BMI, years post-menopause and parity. Pre-procedural data will record history of gynaecological surgery including minor procedures, risk factors for endometrial cancer, medical history, and transvaginal ultrasound scan findings. Intra-procedural data collected for both groups will record whether access to the endometrial cavity was obtained and if not, whether this was due to cervical stenosis or other factors. The contents of the Pipelle® aspiration obtained will be visually assessed by the doctor and if deemed to be an adequate sample this will be sent on for histopathological assessment. In addition, the intervention arm will have intra-procedural data collected to assess whether the Pipelle® was clearly visualised on transabdominal ultrasound and seen at the fundus.

Post-procedural data for both groups will record the number of samples deemed adequate for assessment by the histopathology department and for those not deemed adequate, the specified reason. The histology results will be recorded and the proportion of patients with benign pathology, endometrial hyperplasia (with and without atypia) and endometrial cancer recorded. Any complications occurring during or post procedure will be recorded. Patients will be monitored for repeat attendances during the study, to ensure that any patient later diagnosed with higher order pathology has this recorded.

WITHDRAWAL CRITERIA Patients enrolled in the trial will be free to withdraw consent at any point without giving reason for doing so. If this occurs their care will be returned to standard practice. If the doctor performing the procedure feels at any point it is not safe to proceed, or it is no longer in the patient's best interests, then the procedure will be abandoned and a discussion had as to how best investigate or treat their post-menopausal bleeding. Any decision and reason to withdraw from the study will be recorded.

ASSESSMENT AND FOLLOW-UP Follow up for all trial participants will be the same as for patients undergoing standard assessment of post-menopausal bleeding. Histopathology results will be reviewed within two weeks of the sample being taken and if benign the patient will be discharged from the clinic. Their GP will receive a letter stating that their investigations are normal and their involvement in the trial has come to an end. If they have further episodes of post-menopausal bleeding their GP will be asked to refer them back to the rapid access clinic on a suspected cancer pathway. If non-benign pathology is found, then the patient will be invited for a further appointment and follow up will be determined as per the relevant protocol. If the laboratory reports that the sample taken is not adequate for histopathological analysis the patient will be contacted and recommended to undergo a hysteroscopy for further assessment.

ETHICS APPROVAL The Study Coordination Centre has obtained approval from the London-London Bridge Research Ethics Committee (REC) and Health Research Authority (HRA). The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Helsinki 1964 and later revisions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with post-menopausal bleeding who require an endometrial biopsy.

Further details:

* Post-menopausal bleeding is defined as bleeding one year after a woman's last menstrual period or bleeding six months after starting continuous combined hormone replacement therapy.
* There is no upper age limit, however all patients must be 18 or above.

Strict ultrasound criteria will be followed:

* Endometrium ≥5mm: this is the current cut off used by Imperial College Healthcare NHS Trust for a biopsy to be indicated in the context of post-menopausal bleeding.
* Smooth, homogenous endometrium with a clearly defined border.

Exclusion Criteria:

* Focal endometrial pathology (including but not limited to endometrial polyps, type 0-2 fibroids, uterine septa and other uterine structural abnormalities).
* Suspicion of non-benign myometrial pathology.
* History of endometrial cancer or endometrial hyperplasia.
* History of cervical cancer.
* Virgo intacta.
* Inability to tolerate vaginal examination.
* Inability to consent.
* The denial or withdrawal of informed written consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-07-23 (Estimated); Primary Completion 2027-07-23 (Estimated); Study Completion 2027-07-23 (Estimated)

PRIMARY OUTCOMES:
Adequate endometrial biopsy (Yes/No). | 3 years
  Sufficient intact endometrial tissue to safely diagnose or exclude endometrial cancer and endometrial hyperplasia, as assessed by a histopathologist.

SECONDARY OUTCOMES:
Patient satisfaction (Visual Analogue Scale, 0-10). | 3 years
  Questionnaire with four questions:
  1. What was your level of anxiety leading up to your appointment today? (Visual Analogue Scale showing all numbers 0 - 10, 0 lowest anxiety - 10 highest anxiety)
  2. What was your pain level during your biopsy today? (Visual Analogue Scale showing all numbers 0 - 10, 0 lowest pain - 10 highest pain)
  3. What was your pain level after your biopsy today? (Visual Analogue Scale showing all numbers 0 - 10, 0 lowest pain - 10 highest pain)
  4. How satisfied are you with your experience in the clinic today? (Visual Analogue Scale showing all numbers 0 - 10, 0 lowest satisfaction - 10 highest satisfaction)
Time to treatment (Days). To determine whether women undergoing an outpatient Pipelle® endometrial biopsy performed under transabdominal ultrasound guidance have a shorter time from their biopsy to receiving definitive treatment. | 3 years
  Days from the initial Pipelle® endometrial biopsy attempt until treatment in cases of endometrial cancer or endometrial hyperplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Yazbek, MD, Principal Investigator — Imperial College Healthcare Trust
Locations (1):
- Queen Charlotte's and Chelsea Hospital, Imperial College Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It will not be necessary to share individual participant data (IPD) with other researchers outside of the immediate research team. The only members with access to the information will be the Principal Investigator (Joseph Yazbek) and the study Co-ordinator (Nicholas Anson).